CLINICAL TRIAL: NCT00374270
Title: Improving Blood Pressure Management in Patients With Diabetes: SCRIP-HTN
Brief Title: Improving Blood Pressure Management in Patients With Diabetes
Acronym: SCRIP-HTN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Diabetes Association (Other); Heart and Stroke Foundation of Canada (Other); College and Association of Registered Nurses of Alberta (Other); Alberta Health & Wellness (Other Government); Medicine Shoppe of Canada (Unknown); Canadian Council of Cardiovascular Nurses (Other); MED Institute, Incorporated (Industry); Capital Health, Canada (Other); Alberta Heritage Foundation for Medical Research (Other); Alberta Medical Association (Other); Merck Frosst Canada Ltd. (Industry)
Responsible Party: Dr. Ross Tsuyuki, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EPICORE-GG5130000107
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Hypertension; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes (type I and type II)
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Lifestyle Counselling; Opinion Leader Influence Statements

SUMMARY:
About 22% of Canadians have high blood pressure, or hypertension. However, studies have shown that only 1 out of 5 people with hypertension have their blood pressure controlled.

Diabetes is also an important risk factor for heart disease and stroke. About half of people with diabetes also have hypertension - a deadly combination. Studies have shown that only about 1 in 10 people with diabetes have their blood pressure controlled adequately - clearly something needs to be done to improve this.

Heart disease, stroke, hypertension, and diabetes are conditions that occur in the community, so we need to explore innovative solutions that will work in the community. Pharmacists are well-placed in the community to help identify people with diabetes and hypertension. This has worked very well in previous studies in patients with high cholesterol levels. Pharmacists and nurses have complementary skills which, when working as a team, may help identify and better manage hypertension in people with diabetes.

Our main objective is to test whether a community pharmacist and nurse team can improve blood pressure control in people with diabetes and hypertension.

DETAILED DESCRIPTION:
Background: Cardiovascular disease (CVD) is the leading cause of mortality in Canada. Diabetes is a strong risk factor for CVD, accounting for 50%-75% of deaths (1). Almost half of patients with diabetes also have hypertension. Recent evidence suggests that blood pressure (BP) control is a more important target than blood glucose for the prevention of complications of diabetes, because reducing BP reduces the risks of both CVD and renal dysfunction (2-4). Despite this, and recommendations from national guidelines, BP control in individuals with diabetes is poor (5-10). We recently performed a systematic review of 43 studies, (72,237 patients), and observed that only about 40% achieve treatment targets (11). This is likely an overestimate, as all studies used BP targets higher than current recommendations. Community pharmacists and advanced nurse practitioners (ANP) are well-positioned to help identify and follow-up patients with diabetes and hypertension.

Objective: To determine the efficacy of a community-based multidisciplinary screening and intervention program on blood pressure control in patients with diabetes.

Design and Methods: Design: Subjects will be randomized to pharmacist/ANP intervention or usual care. Inclusion criteria: Adult patients with diabetes with a BP of >130/80 mm Hg on 2 consecutive visits 2 weeks apart. Exclusion criteria: patients who are institutionalized or unlikely/unable to comply with follow up visits. Procedures: Patients will be recruited via: 1) community pharmacies (patients identified by diabetes drug prescriptions), and 2) referrals via Capital Health Regional Diabetes Intake Program. Patients will be invited by telephone to attend an in-pharmacy clinic. At Visit #1, the ANP will complete a history and physical exam (including a BP taken using the BPTru® device, 6 readings performed 1 minutes apart in the non-dominant arm, with last 5 readings averaged) (12). The pharmacist will review each patient's medication history. If the averaged readings are >130/80 mm Hg, the patient will be invited to attend a 2nd clinic in 2 weeks. If the averaged BPs from both visits are >130/80 mm Hg, the patient will be approached for consent to participate in the randomized trial. Intervention group receives: a BP wallet card with discussion as to the meaning of the BP measures, CVD risk reduction counseling, a hypertension education pamphlet, and referral to their primary care physician for further assessment/management. The BP results will then be faxed along with any recommendations to the patient's primary care physician. Written recommendations from local opinion leaders will be used to reinforce the latest hypertension guidelines. Follow-up: Patients will be followed up at 6 weeks to ensure they have made an appointment with their physician and to re-measure BP. BP will be measured at 6-week intervals (Week 6, 12, 18 with faxing of BP results and recommendations to the primary care physician), with a final follow-up visit at Week 24. Usual care group receives: BP wallet card with recorded BP measures, a pamphlet on diabetes, general diabetes advice given by ANP and usual care by their physician. Follow-up: No scheduled follow up visits. One phone call to patient will occur at 12 weeks to inquire about changes to BP management. A final follow-up visit will occur at week 24 to re-evaluate BP and to offer the patients the intervention program.

Evaluation: Outcome measures: The primary endpoint is the difference in change in systolic BP between intervention and usual care groups at 6 months. Secondary endpoints will include: (1) change in antihypertensive therapy (new medication or dosage increase), (2) % patients achieving BP target of <130/80 mm Hg, and (3) % patients using ACE inhibitors or angiotensin receptor antagonists. Sample Size: A sample size of 85 patients per group will provide 90% power (assuming a standard deviation of 20mmHg and 2-sided alpha=0.05) to detect a 10mmHg difference in the primary endpoint. To account for drop-outs, we will increase this to 110 patients per group. Analysis: Demographic characteristics will be summarized using percentages for categorical variables and medians (interquartile range) for continuous variables. To compare the change in BP between intervention and usual care, we will use a 2-sample independent t-test. Significance of Study: Treatment and control of hypertension in people with diabetes is a major public health problem, and improving detection and control of hypertension is a major goal of the Canadian Hypertension Society. Novel ways of identification and treatment to guideline targets in this patient population are urgently needed.

ELIGIBILITY:
Inclusion Criteria:

The following patients will be eligible for study participation:

* Patients with either type 1 or type 2 diabetes. Diabetes will be defined as those patients presently taking either oral hypoglycemic agents or insulin therapy (oral hypoglycemic agents to include all drugs in the drug classes of: alpha-glucosidase inhibitors, biguanides, meglitinides, sulfonylureas, thiazolidinediones and adjunctive therapy) taken for >6 months to rule-out steroid-induced diabetes and gestational diabetes.

Exclusion Criteria:

Patients will be excluded from the study if they:

* Do not provide or are unable to provide written informed consent
* Refuse or are unlikely to attend follow-up visits for BP measurements
* Are institutionalized
* Are <18 years of age
* Do not understand English
* Enrolled in other diabetes or hypertension trials

Subjects will be recruited whether or not they are receiving antihypertensive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2005-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
difference in change in systolic BP between the intervention and usual care groups | 6 months

SECONDARY OUTCOMES:
change in antihypertensive therapy by new/additional hypertension medication or dosage increase between groups | 6 months
proportion of patients achieving goal BP of <130/80 mm Hg between groups | 6 months
proportion of patients that are prescribed an ACE inhibitor or angiotensin receptor antagonist between groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ross T Tsuyuki, PharmD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] McLean DL, McAlister FA, Johnson JA, King KM, Makowsky MJ, Jones CA, Tsuyuki RT; SCRIP-HTN Investigators. A randomized trial of the effect of community pharmacist and nurse care on improving blood pressure management in patients with diabetes mellitus: study of cardiovascular risk intervention by pharmacists-hypertension (SCRIP-HTN). Arch Intern Med. 2008 Nov 24;168(21):2355-61. doi: 10.1001/archinte.168.21.2355. PMID 19029501
- See also: Related Info — https://www.epicore.ualberta.ca